CLINICAL TRIAL: NCT00000893
Title: A Phase I/II, Open-Label, AUC-Controlled Study to Determine the Pharmacokinetics, Safety, Tolerability, and Antiviral Activity of DMP 266 (Efavirenz) in Combination With Nelfinavir in Children
Brief Title: Safety, Tolerability, and Anti-HIV Activity of DMP 266 (Efavirenz) in Combination With Nelfinavir in HIV-Positive Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 382; 10105 (Registry Identifier: DAIDS ES); PACTG 382
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Drug Therapy, Combination; HIV Protease Inhibitors; Nelfinavir; Reverse Transcriptase Inhibitors; Area Under Curve; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Nelfinavir; efavirenz

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Efavirenz

SUMMARY:
Cohort I: The purpose of this study is to see how safe it is to combine 2 anti-HIV medications, efavirenz (EFZ) and nelfinavir (NFV) to treat HIV-positive children and to find an appropriate dose of EFZ to use in combination with NFV. Cohort II: The purpose of this study is to see how safe it is to give EFZ syrup combined with NFV and to measure the levels of EFZ and NFV in the blood. (This purpose reflects a change from the original since there are now 2 different cohorts of patients.) EFZ is an effective anti-HIV medication that easily can be combined with other drugs to treat HIV. This is an early study to determine a safe and effective dose for HIV-positive children. This study also will examine the correct dose of NFV to use in combination with EFZ.

DETAILED DESCRIPTION:
The demonstrated antiviral activity, tolerability, and pharmacokinetic properties of DMP 266 and its utility in combination with other agents make DMP 266 an attractive agent for use in HIV-infected pediatric patients. However, the tolerability of DMP 266 in the pediatric population must be evaluated, and appropriate dosing instructions need to be developed. By following the patients over time, the antiviral activity of DMP 266-containing regimens will be documented. Dosage guidelines for children can then be developed following analysis of the results.

This is a 48-week [AS PER AMENDMENT (APA) 12/21/98:104-week] [APA 5/8/00: 208-week] study. It is designed to minimize the chance that ineffective therapy is provided (short dose-escalation phase) and utilizes an area under the concentration time curve (AUC) to establish plasma levels of DMP 266 and nelfinavir in the pediatric population that are both tolerable and efficacious. [APA 5/26/98: Patients are stratified by age into Cohorts I and II] and receive EFV concurrently with NFV.

[APA 5/26/98: The initial starting dose of DMP 266 for patients in Cohort II is higher than the initial starting dose for patients in Cohort I.] [APA 12/21/98: The initial starting dose for patients in Stratum 1 of Cohort II is higher than the initial starting dose for patients in Cohort I and Stratum 2 of Cohort II.] The initial target AUC for DMP 266 is between 190 and 380 micromoles/h (uM/h). The initial starting dose (based on a 70 kg patient and adjusted for each patient's weight) for the first 6 patients is adjusted on the basis of tolerability and plasma concentrations of DMP 266 after 2 weeks of daily doses. If at least 4 of the first 6 patients attain a tolerable dose (dose at which no more than 2 of 6 patients experience Grade 3 or worse toxicity) and target AUC, additional patients may continue to be accrued. However, if any of the initial 6 patients experience life-threatening toxicity, further accrual is suspended. [APA 5/26/98: An assessment of the tolerability and plasma concentrations of EFV is not required in an initial group of Cohort II patients. Individual dose is based on pharmacokinetic sampling.] Patients receive a given starting dose of DMP 266 and continue on that dose until individual dose adjustments are needed. If a patient's starting dose is tolerated but the target AUC is not achieved, the dose is increased. If the starting dose is well tolerated and target AUC achieved, no adjustment in starting dose is given to future patients. If no tolerated dose achieving at least an AUC of 150 micromoles/h is reached in 4 of 6 patients, the study is suspended and alternative dosing regimens, e.g., twice-daily dosing, are considered.

A patient's current dose of DMP 266 is adjusted based on how the dose is tolerated and whether the target AUC is achieved. If a patient does not achieve an AUC of greater than 110 micromoles/h and experiences Grade 3 or worse toxicity, the patient is discontinued from the study.

[APA 12/21/98: The dose of NFV is the same for patients in Cohort I and Stratum 2 of Cohort II; the dose for patients in Stratum 1 of Cohort II is higher.] The minimum target AUC for NFV is 10 mg x h/L. Doses are adjusted for an individual child if AUC falls below threshold at Week 2 or 6. Children with weight no greater than 30 kg receive a lower dose than children with weight greater than 30 kg or Tanner Stage IV. [APA 5/8/00: The first group of 6 patients receives the initial dose of NFV. If none of the 6 patients falls below the target AUC, the remainder of the sample is accrued and treated at this dose. If more than 1 of the 6 patients fall below the target AUC, then another group of 6 patients is accrued and treated at the next higher dose. If exactly 1 of the 6 patients falls below the target AUC, 2 more patients are accrued and treated at the same dose. If 1 of these 2 patients falls below the target AUC, another group of 6 patients is tested on the next higher dose. If neither of these 2 patients falls below the target AUC, then the remainder of the sample is accrued and treated at this dose. The dose is escalated until a dose that meets the above criteria is achieved or further dose escalation is prohibited due to toxicity.] The duration of therapy is 48 [APA 12/21/98:104] [APA 5/8/00: 208] weeks.

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are HIV-positive.
* Are between 3 months and 16 years old (consent of parent or legal guardian required). (These age requirements reflect a change.)
* Have a plasma viral load of at least 400 copies/ml at screening.
* Agree to practice abstinence or use effective methods of birth control during the study.
* Are able to take oral medication and comply with study requirements.
* Are taking at least 1 nucleoside reverse transcriptase inhibitor (NRTI), such as zidovudine (ZDV) or stavudine (d4T). Patients can begin taking NRTIs at the beginning of the study.

Exclusion Criteria

Children will not be eligible for this study if they:

* Have had more than 2 episodes of moderate to severe diarrhea or vomiting lasting more than 4 days within 3 months prior to study entry.
* Are allergic to EFZ or NFV.
* Have any disease, including hepatitis, cancer, or an active opportunistic (HIV-associated) infection.
* Are pregnant or breast-feeding.
* Are taking any other experimental drugs or certain medications.
* Have ever taken protease inhibitors (PIs) or nonnucleoside reverse transcriptase inhibitors (NNRTIs).

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 1997-10; Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Fletcher, Study Chair; Stuart Starr, Study Chair
Locations (27):
- United States (25):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Usc La Nichd Crs, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Univ. of Mississippi Med. Ctr Children's Hosp., Jackson, Mississippi
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - Metropolitan Hosp. Ctr., New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Nyu Ny Nichd Crs, New York, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Texas Children's Hosp. CRS, Houston, Texas
  - Seattle Children's Hospital CRS, Seattle, Washington
  - UW School of Medicine - CHRMC, Seattle, Washington
- Puerto Rico (2):
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Brundage RC, Fletcher CV, Fiske WD, Kornhauser DM, McNamara J, Mofenson L, Starr SE. Pharmacokinetics of an efavirenz suspension in children. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:147 (abstract no 424)
- [Background] Fletcher CV, Fenton T, Powell C, Anderson PL, Brundage RC, Spector SA, Starr SE. Pharmacologic characteristics of efavirenz (EFV) and nelfinavir (NFV) associated with virologic response in HIV-infected children. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 259)
- [Background] Saitoh A, Hsia K, Fenton T, Powell C, Christopherson C, Fletcher CV, Starr SE, Spector SA. HIV-1 DNA persists in PBMC of children on HAART despite prolonged suppression of plasma HIV-1 RNA. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 685B)
- [Background] Fletcher CV, Brundage RC, Fenton T, Fiske WD, Kornhauser D, McNamara J, Mofenson L, Starr SE. Efavirenz (EFV) and nelfinavir (NFV) pharmacokinetics (PK) in HIV-infected children participating in an area under the curve (AUC) controlled trial. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:136 (abstract no 366)
- [Result] Starr SE, Fletcher CV, Spector SA, Yong FH, Fenton T, Brundage RC, Manion D, Ruiz N, Gersten M, Becker M, McNamara J, Mofenson LM, Purdue L, Siminski S, Graham B, Kornhauser DM, Fiske W, Vincent C, Lischner HW, Dankner WM, Flynn PM. Combination therapy with efavirenz, nelfinavir, and nucleoside reverse-transcriptase inhibitors in children infected with human immunodeficiency virus type 1. Pediatric AIDS Clinical Trials Group 382 Team. N Engl J Med. 1999 Dec 16;341(25):1874-81. doi: 10.1056/NEJM199912163412502. PMID 10601506
- [Result] Spector SA, Hsia K, Yong FH, Cabral S, Fenton T, Fletcher CV, McNamara J, Mofenson LM, Starr SE. Patterns of plasma human immunodeficiency virus type 1 RNA response to highly active antiretroviral therapy in infected children. J Infect Dis. 2000 Dec;182(6):1769-73. doi: 10.1086/317621. Epub 2000 Oct 26. PMID 11069252
- [Result] Saitoh A, Singh KK, Powell CA, Fenton T, Fletcher CV, Brundage R, Starr S, Spector SA. An MDR1-3435 variant is associated with higher plasma nelfinavir levels and more rapid virologic response in HIV-1 infected children. AIDS. 2005 Mar 4;19(4):371-80. doi: 10.1097/01.aids.0000161766.13782.2f. PMID 15750390
- [Result] Saitoh A, Fenton T, Alvero C, Fletcher CV, Spector SA. Impact of nucleoside reverse transcriptase inhibitors on mitochondria in human immunodeficiency virus type 1-infected children receiving highly active antiretroviral therapy. Antimicrob Agents Chemother. 2007 Dec;51(12):4236-42. doi: 10.1128/AAC.00893-07. Epub 2007 Sep 24. PMID 17893156